CLINICAL TRIAL: NCT01526694
Title: Phase II Multicenter Clinical Trial to Investigate the Efficacy and Safety of Bendamustine, Dexamethasone and Thalidomide in R/R MM Pts After Treatment With Lenalidomide and Bortezomib or Which Are Ineligible to One of These Drugs
Brief Title: Phase II Trial Designed to Determine Efficacy and Safety of Bendamustine+Dexamethasone+Thalidomide in R/R MM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Azienda Ospedaliera di Bolzano (Other)
Collaborators: Mundipharma Pte Ltd. (Industry)
Responsible Party: Principal Investigator, Michael Mian, MD, Azienda Ospedaliera di Bolzano
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BDT-01-2011
Record Dates: First submitted 2012-01-27; First posted 2012-02-06 (Estimated); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Multiple Myeloma
Keywords: relapsed or refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — Bendamustine Hydrochloride; Thalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- treatment with BDT (Experimental): Bendamustine + Dexamethasone + Thalidomide in patients with multiple myeloma (MM) patients after treatment with lenalidomide and bortezomib or which are ineligible to one of these drugs.
  Interventions: Drug: Bendamustine; Drug: Thalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Bendamustine — Bifunctional alkylating agent consisting of a purine and amino acid antagonist (a benzimidazole ring) and an alkylating nitrogen mustard moiety.
  Other Names: Ribomustin
Drug: Thalidomide — Thalidomide can directly inhibit the growth and survival of myeloma cells, by oxidative damage to DNA mediated by free radicals. The drug can induce apoptosis even in drug resistant myeloma cells. Thalidomide modulates cell adhesion molecule expression, so it may interfere with the mutually stimulatory interactions between myeloma cells and the bone marrow microenvironment.
Drug: Dexamethasone — It's a corticosteroid.

SUMMARY:
This is a prospective, multicenter phase II trial designed to determine efficacy and safety of a combination chemotherapy consisting of Bendamustine + Dexamethasone + Thalidomide in patients with multiple myeloma (MM) after treatment with lenalidomide and bortezomib or which are ineligible to one of these drugs.

DETAILED DESCRIPTION:
Eligible patients will be treated according to the following scheme until the occurrence of maximum response, dose limiting toxicity or disease progression. Repeat cycles every 28 days for a maximum of 6 cycles and a minimum of 4.

* Bendamustine 60 mg/m2 i.v. days 1, 8, 15
* Dexamethasone 20 mg p.o. days 1,8 , 15, 22
* Thalidomide 100 mg daily p.o. days 1-28; initial dose of 50 mg/day, with an increment to 100 mg after the first 15 days of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent form.
* Age 18 years at the time of signing the informed consent form.
* Life expectancy of at least 3 months
* Able to adhere to the study visit schedule and other protocol requirements
* Relapsed or refractory active MM (according to the International Myeloma Working Group guidelines) after treatments containing bortezomib and lenalidomide or ineligible (intolerance or toxicity) to one of these drugs with detectable myeloma protein in blood or urine.
* Disease free of prior malignancies for at least 5 years.
* All previous multiple myeloma treatments, including radiation, cytostatic therapy and surgery, must have been discontinued at least 4 weeks prior to treatment in this study, except corticosteroids therapy.
* ECOG performance status <2 at study entry, unless it is due to MM.
* At least the following laboratory findings at the day of treatment start:
* Platelet count ≥ 75 x 10^9/L without transfusional support within 7 days.
* Neutrophil count > 1.5 x 10^9/L without G-CSF.
* Corrected calcium ≤ 14 mg/dL (3.5 mmol/L).
* AST: ≤ 2.5 times the normal upper limit.
* ALT: ≤ 2.5 times the normal upper limit.
* Total bilirubin: ≤ 1.5 times the normal upper limit.
* Measured or calculated creatinine clearance of ≥ 20 mL/minute
* Women of child bearing potential and male patients whose partner is a woman of child bearing potential must be prepared to use two effective methods of contraception both before and during protocol treatment, or commit to absolute and continuous abstinence.The pregnancy test must be negative 14-28 days and 72 hours before treatment start. Only in case of hysterectomy or presence of menopause for at least 24 consecutive months pregnancy tests as well as contraception are not necessary. Men must not father a child for up to 6 months following cessation of treatment and must use condoms.

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Pregnant or breast feeding females.
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Patients with contraindications for treatment with bendamustine, dexamethasone and thalidomide.
* Uncontrolled or severe cardiovascular disease, including myocardial infarction within 6 months before study entry, New York Heart Association Class III or IV heart failure, uncontrolled angina or severe uncontrolled ventricular arrhythmias (≥ Lown 3).
* Use of any other experimental drug or therapy within 28 days of baseline.
* Known hypersensitivity to thalidomide or purine analogues
* Concurrent use of other anti-cancer agents or treatments other stated in this treatment plan.
* Peripheral neuropathy grade ≥2 according to WHO
* Known positive for HIV or infectious hepatitis, type A, B or C.
* Major surgery less than 30 days before start of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2017-04-08 (Actual)

PRIMARY OUTCOMES:
Response rate | 18 months
  The proportion of patient with a Complete Response (CR) or Very Good Partial Response or partial response
Incidence of haematological toxicity of BDT | 18 months
  The incidence of haematological toxicities is the proportion of patients with haematological toxicity

SECONDARY OUTCOMES:
Time to treatment Failure (TTF) | 18 months
  To evaluate time to treatment failure
Survival (OS) | 18 months
  To evaluate overall survival
Disease Free Survival (DFS) | 18 months
  To evaluate disease free survival

CONTACTS AND LOCATIONS:
Overall Officials: Michael Mian, MD, Principal Investigator — Azienda Ospedaliera di Bolzano
Locations (19):
- Italy (19):
  - Division of Hematology and CBMT, Bolzano, BZ
  - Presidio Ospedaliero di Camposampiero, Camposampiero, Padova
  - Ospedale S. Martino, Belluno
  - Ospedale di Castelfranco Veneto, Castelfranco Veneto
  - Ospedale Civile di Dolo, Dolo
  - AULSS 2 Feltre, Feltre
  - Azienda Ospedaliera Universitaria G. Martino, Messina
  - Ospedale dell'Angelo di Mestre, Mestre
  - A.O di Padova Ematologia e Immunologia Clinica, Padua
  - A.O di Padova Ematologia, Padua
  - AULLS 18 di Rovigo, Rovigo
  - Ospedale di Trento - P.O. S. Chiara, Trento
  - Ospedale Ca Foncello, Treviso
  - A.O.U Ospedali Riuniti di Trieste Medicina II, Trieste
  - A.O.U Ospedali Riuniti di Trieste, Trieste
  - A.O.U S. Maria della Misericordia, Udine
  - Ospedale Policlinico G.B Rossi (Borgo Roma) Ematologia, Verona
  - Ospedale Policlinico G.B Rossi (Borgo Roma) Medicina II, Verona
  - AULSS 6 Vicenza, Vicenza

IPD SHARING:
Plan to Share IPD: No